CLINICAL TRIAL: NCT01816971
Title: Phase 2 Study of the Initial and Post-Transplant Treatment With Carfilzomib, Lenalidomide and Low Dose Dexamethasone (CRd) in Transplant Candidates With Newly Diagnosed, Multiple Myeloma Requiring Systemic Chemotherapy
Brief Title: Carfilzomib, Lenalidomide, and Dexamethasone Before and After Stem Cell Transplant in Treating Patients With Newly Diagnosed Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-1725; NCI-2012-02023 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Results first posted 2022-09-23 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Dexamethasone; Calcium Dobesilate; carfilzomib; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (dexamethasone, carfilzomib, lenalidomide) (Experimental): INDUCTION THERAPY: Patients receive dexamethasone IV or PO QD on days 1, 8, 15 and 22; carfilzomib IV over 10-30 minutes on days 1, 2, 8, 9, 15, and 16; and lenalidomide PO QD on days 1-21. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity..
  TRANSPLANT: Patients undergo autologous stem cell transplant.
  CONSOLIDATION THERAPY: Patients receive dexamethasone, carfilzomib, and lenalidomide as in induction. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive dexamethasone and lenalidomide as in induction therapy and carfilzomib IV over 30 minutes on days 1, 2, 15, and 16. Treatment repeats every 28 days for 10 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: dexamethasone; Drug: carfilzomib; Drug: lenalidomide; Procedure: autologous hematopoietic stem cell transplantation; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: dexamethasone — Given IV or PO
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM
Drug: carfilzomib — Given IV
  Other Names: Kyprolis; PR-171
Drug: lenalidomide — Given PO
  Other Names: CC-5013; IMiD-1; Revlimid
Procedure: autologous hematopoietic stem cell transplantation — Undergo autologous hematopoietic stem cell transplant
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well carfilzomib, lenalidomide, and dexamethasone before and after stem cell transplant works in treating patients with newly diagnosed multiple myeloma. Carfilzomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Biological therapies, such as lenalidomide, may stimulate the immune system in different ways and stop cancer cells from growing. Drugs used in chemotherapy, such as dexamethasone, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from diving. Giving carfilzomib, lenalidomide, and dexamethasone before and after stem cell transplant may kill more cancer cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the rate of stringent complete response (CR) (sCR) after 8 cycles of CRd (4 cycles of induction + autologous stem cell transplant [ASCT] + 4 cycles of carfilzomib, lenalidomide, and low dose dexamethasone [CRd] consolidation).

SECONDARY OBJECTIVES:

I. Overall response rate defined as partial response or better (>= partial response [PR]) including the rate of very good partial response (VGPR) or better (>= VGPR) and near complete response or better (sCR/CR/nCR) across entire treatment in high risk and low risk patients.

II. Duration of response (DOR), progression free survival (PFS), time to progression (TTP), and overall survival (OS).

TERTIARY OBJECTIVES:

I. Determination of the rate of minimal residual disease in patients who achieved CR.

II. Prospective evaluation of candidate markers of response to CRd established in the completed CRd trial.

III. Evaluation of markers of response and duration of response to treatment strategy using CRd with or without transplant.

OUTLINE:

INDUCTION THERAPY: Patients receive dexamethasone intravenously (IV) or orally (PO) once daily (QD) on days 1, 8, 15 and 22; carfilzomib IV over 10-30 minutes on days 1, 2, 8, 9, 15, and 16; and lenalidomide PO QD on days 1-21. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity..

TRANSPLANT: Patients undergo autologous stem cell transplant.

CONSOLIDATION THERAPY: Patients receive dexamethasone, carfilzomib, and lenalidomide as in induction. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Patients receive dexamethasone and lenalidomide as in induction therapy and carfilzomib IV over 30 minutes on days 1, 2, 15, and 16. Treatment repeats every 28 days for 10 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, myeloma requiring systemic chemotherapy as per International Myeloma Working Group (IMWG) uniform criteria:

  * Prior treatment of hypercalcemia or spinal cord compression or active and/or aggressively progressing myeloma with corticosteroids or lenalidomide or bortezomib-based regimens does not disqualify the patient (the treatment dose should not exceed the equivalent of 160 mg of dexamethasone in a 4 week period or not more than 1 cycle)
  * Bisphosphonates are permitted
* Suitable and interested to proceed to ASCT
* Measurable disease, prior to initial treatment as indicated by one or more of the following:

  * Serum monoclonal (M)-protein >= 0.5 g/dL
  * Urine M-protein >= 200 mg/24 hours
  * If serum protein electrophoresis is felt to be unreliable for routine M-protein measurement, then quantitative immunoglobulin levels are acceptable
* Life expectancy of more than 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Bilirubin < 1.5 times the upper limit of normal (ULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 times ULN
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L
* Hemoglobin >= 8 g/dL
* Platelet count >= 75 x 10^9/L; subjects may receive red blood cell (RBC) transfusions or platelet transfusions, if clinically indicated in accordance with institutional guidelines; however, screening platelet count should be independent of platelet transfusions for at least 2 weeks
* Calculated or measured creatinine clearance of >= 50 mL/minute, calculated using the formula of Cockcroft and Gault
* Written informed consent in accordance with federal, local, and institutional guidelines
* Females of childbearing potential (FCBP) (defined as sexually mature females who: have not undergone a hysterectomy or bilateral oophorectomy; or have not been naturally postmenopausal for at least 24 consecutive months [ie, has had menses at any time in the preceding 24 consecutive months]) must agree to ongoing pregnancy testing
* FCBP must have 2 negative pregnancy tests (sensitivity of at least 50 mIU/mL) prior to initiating lenalidomide; the first pregnancy test must be performed within 10-14 days before day 1 cycle 1 and the second pregnancy test must be performed within 24 hours of day 1 cycle 1; the subject may not receive lenalidomide until the treating investigator has verified that the results of these pregnancy tests are negative, and must agree to ongoing pregnancy tests as outlined in the protocol
* FCBP must agree to use 2 reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual intercourse during the following time periods related to this study:

  * For at least 28 days before starting lenalidomide
  * While participating in the study; and
  * For at least 28 days after discontinuation from the study; the 2 methods of reliable contraception must include a highly effective method (ie, intrauterine device (IUD), hormonal [birth control pills, injections, or implants], tubal ligation, partner's vasectomy) and an additional effective (barrier) method (ie, latex condom, diaphragm, cervical cap); FCBP must be referred to a qualified provider of contraceptive methods if needed
* Male subjects must agree to use a latex condom during sexual contact with females of childbearing potential while participating in the study and for at least 28 days following discontinuation from the study even if he has undergone a successful vasectomy
* Male subjects must agree to inform his physician if he has had unprotected sexual contact with a female who can become pregnant or if he thinks for any reason that his sexual partner may be pregnant
* Male subjects must agree not to donate semen or sperm while taking lenalidomide
* All study participants must be registered into the mandatory Rev Assist program and be willing and able to comply with the requirements of Rev Assist
* The ability to take aspirin or other appropriate venous thromboembolism (VTE) prophylaxis
* Subjects must agree to adhere to all study requirements, including birth control measures and pregnancy testing, visit schedule, outpatient treatment, required concomitant medications, and laboratory monitoring

Exclusion Criteria:

* Non-secretory or hyposecretory multiple myeloma, prior to initial treatment defined as < 0.5 g/dL M-protein in serum, < 200 mg/24 hr urine M-protein, or disease only measured by serum free light chain
* POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
* Waldenstrom's macroglobulinemia or immunoglobin (Ig)M myeloma
* Radiotherapy to multiple sites or immunotherapy within 4 weeks before start of protocol treatment (localized radiotherapy to a single site at least 1 week before start is permissible)
* Participation in an investigational therapeutic study within 3 weeks or within 5 drug half-lives (t1/2) prior to first dose, whichever time is greater
* Pregnant or lactating females
* History of allergy to mannitol
* Major surgery within 3 weeks prior to first dose
* Myocardial infarction within 6 months prior to enrollment, New York Heart Association (NYHA) class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Uncontrolled hypertension or diabetes
* Acute active infection requiring systemic antibiotics, antivirals, or antifungals within two weeks prior to first dose
* Known or suspected human immunodeficiency virus (HIV) infection, known HIV seropositivity
* Active hepatitis A, B, or C infection
* Non-hematologic malignancy within the past 3 years except adequately treated basal cell, squamous cell skin cancer, thyroid cancer, carcinoma in situ of the cervix, or prostate cancer < Gleason grade 6 with stable prostate specific antigen levels or cancer considered cured by surgical resection alone
* Any clinically significant medical disease or condition that, in the investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent
* Significant neuropathy (grades 3-4, or grade 2 with pain) at the time of the first dose and/or within 14 days before enrollment
* Contraindication to any of the required concomitant drugs, including proton-pump inhibitor (eg, lansoprazole), enteric-coated aspirin, allopurinol or if a history of prior thrombotic disease, warfarin or low molecular weight heparin
* Subjects in whom the required program of PO and IV fluid hydration is contraindicated, eg, due to pre-existing pulmonary, cardiac, or renal impairment
* Subjects with known or suspected amyloidosis of any organ
* Subjects with pleural effusions requiring thoracentesis or ascites requiring paracentesis
* No coverage or not-acceptable by patient co-pay for lenalidomide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-01; Primary Completion 2018-04-01 (Actual); Study Completion 2026-12-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Andrzej Jakubowiak, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (5):
- United States (4):
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Dana Farber, Boston, Massachusetts
  - Washington University in St Louis, St Louis, Missouri
  - Sarah Cannon Cancer Center, Nashville, Tennessee
- Princess Margaret, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Landgren O, Kazandjian D, Roussel M, Jasielec J, Dytfeld D, Anderson A, Kervin TA, Iskander K, McFadden I, Jakubowiak AJ. Efficacy and safety of carfilzomib-lenalidomide-dexamethasone in newly diagnosed multiple myeloma: pooled analysis of four single-arm studies. Leuk Lymphoma. 2022 Oct;63(10):2413-2421. doi: 10.1080/10428194.2022.2068001. Epub 2022 May 12. PMID 35549810
- [Derived] Jasielec JK, Kubicki T, Raje N, Vij R, Reece D, Berdeja J, Derman BA, Rosenbaum CA, Richardson P, Gurbuxani S, Major S, Wolfe B, Stefka AT, Stephens L, Tinari KM, Hycner T, Rojek AE, Dytfeld D, Griffith KA, Zimmerman TM, Jakubowiak AJ. Carfilzomib, lenalidomide, and dexamethasone plus transplant in newly diagnosed multiple myeloma. Blood. 2020 Nov 26;136(22):2513-2523. doi: 10.1182/blood.2020007522. PMID 32735641

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Dexamethasone, Carfilzomib, Lenalidomide): INDUCTION THERAPY: Patients receive dexamethasone IV or PO QD on days 1, 8, 15 and 22; carfilzomib IV over 10-30 minutes on days 1, 2, 8, 9, 15, and 16; and lenalidomide PO QD on days 1-21. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity..
  TRANSPLANT: Patients undergo autologous stem cell transplant.
  CONSOLIDATION THERAPY: Patients receive dexamethasone, carfilzomib, and lenalidomide as in induction. Treatment repeats every 28 days for 4 courses in the absence of disease progression or unacceptable toxicity.
  MAINTENANCE THERAPY: Patients receive dexamethasone and lenalidomide as in induction therapy and carfilzomib IV over 30 minutes on days 1, 2, 15, and 16. Treatment repeats every 28 days for 10 courses in the absence of disease progression or unacceptable toxicity.
  dexamethasone: Given IV or PO
  carfilzomib: Given IV
  lenalidomide: Given PO
  autologous hematopoietic stem cell transplantation: Undergo autologous hematopoietic stem cell transplant
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | Treatment (Dexamethasone, Carfilzomib, Lenalidomide)
Started | 76
Completed | 64
Not Completed | 12

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Dexamethasone, Carfilzomib, Lenalidomide)
Number analyzed (Participants) | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 55
  >=65 years | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 59
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 7
  United States | 69

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Achieving sCR
Description: The percentage of stringent complete response (CR) (sCR) will be reported along with 95% confidence intervals, adjusted for the two-stage nature of the trial design.
Time Frame: Day 224
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Dexamethasone, Carfilzomib, Lenalidomide)
Number analyzed (Participants) | 76
percentage of participants | 76 [66 to 84]

2. Secondary Outcome: Overall Response Rate, Defined as at Least a Partial Response to Therapy (> PR), at Least Very Good Partial Response (VGPR) and at Least Near Complete Response (nCR) Rate
Description: Reported along with its exact 95% binomial confidence interval.
Time Frame: Up to 5 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Dexamethasone, Carfilzomib, Lenalidomide)
Number analyzed (Participants) | 76
percentage of participants | 97 [91 to 100]

3. Secondary Outcome: Time to Progression
Description: Estimated using the product-limit method of Kaplan and Meier.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Treatment (Dexamethasone, Carfilzomib, Lenalidomide)
Number analyzed (Participants) | 76
month | NA [NA to NA] — With median follow-up time of 56.0 months, time to progression has not reached the median by the Kaplan-Meier method.

4. Secondary Outcome: Duration of Response
Description: Reported along with its exact 95% binomial confidence interval. Estimated using the product-limit method of Kaplan and Meier.
Time Frame: Up to 5 years
Measure: Median (95% Confidence Interval); unit: month
Arm/Group | Treatment (Dexamethasone, Carfilzomib, Lenalidomide)
Number analyzed (Participants) | 76
month | NA [NA to NA] — With median follow-up time of 56.0 months, duration of response has not reached the median by the Kaplan-Meier method.

5. Secondary Outcome: Percentage of Participants With Progression-free Survival (PFS)
Description: Progression-free Survival rate was estimated at months 12, 24, 36, 48, and 60, by the product-limit method of Kaplan and Meier.
Time Frame: Up to 5 years
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Dexamethasone, Carfilzomib, Lenalidomide)
Number analyzed (Participants) | 76
percentage of participants
  PFS rate at 12 months (%) | 97
  PFS rate at 24 months(%) | 93
  PFS rate at 36 months(%) | 80
  PFS rate at 48 months(%) | 76
  PFS rate at 60 months(%) | 72

6. Secondary Outcome: Percentage of Participants With Overall Survival (OS)
Description: Overall survival rate was estimated at months 12, 24, 36, 48, and 60, by the product-limit method of Kaplan and Meier.
Time Frame: Up to 5 years
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Dexamethasone, Carfilzomib, Lenalidomide)
Number analyzed (Participants) | 76
percentage of participants
  OS rate at 12 months (%) | 100
  OS rate at 24 months (%) | 97
  OS rate at 36 months (%) | 96
  OS rate at 48 months (%) | 93
  OS rate at 60 months (%) | 84

ADVERSE EVENTS:
Time Frame: adverse events (AEs) were collected from the day of treatment initiation through 30 days post-last dose or at the initiation of a new anticancer therapy, up to 5 years.
Description: AEs were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
  Per protocol, AEs were not collected during ASCT (stem cell collection through start of consolidation) and during single-agent lenalidomide maintenance.
Arm/Group | Treatment (Dexamethasone, Carfilzomib, Lenalidomide)
All-Cause Mortality (participants affected / at risk) | 12/76
Serious Adverse Events (participants affected / at risk) | 27/76
Other Adverse Events (participants affected / at risk) | 76/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Dexamethasone, Carfilzomib, Lenalidomide) (N=76)
serious cardiovascular events (Cardiac disorders) | 27 (54)
Fever (General disorders) | 10 (10)
Lung infection (Infections and infestations) | 2 (4)
Non-cardiac chest pain, pleuritic (General disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Eye disorders (Eye disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Flu like symptoms (General disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 3 (3)
Infections and infestations (Infections and infestations) | 1 (1)
Joint infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1)
Burkitt lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Seizure, tonic clonic (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Nervous system disorders (Nervous system disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
shingles outbreak near port-a-cath site (Infections and infestations) | 1 (1)
Thromboembolic Event (Vascular disorders) | 4 (4)
Abdominal Pain (Gastrointestinal disorders) | 1 (2)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin and subcutaneous disorders (Skin and subcutaneous tissue disorders) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1)
Enterocolitis Infection (Infections and infestations) | 1 (1)
ALT Elevation (Investigations) | 1 (1)
colitis (Gastrointestinal disorders) | 1 (1)
Cytokine Release Syndrome (Immune system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Dexamethasone, Carfilzomib, Lenalidomide) (N=76)
Cardiac disorders (Cardiac disorders) | 10 (15)
Thromboembolic events (Vascular disorders) | 14 (15)
Hypertension (Vascular disorders) | 15 (23)
Hypophosphatemia (Metabolism and nutrition disorders) | 22 (49)
Rash (Infections and infestations) | 33 (62)
Peripheral neuropathy (Nervous system disorders) | 32 (41)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 30 (47)
Hyperglycemia (Metabolism and nutrition disorders) | 33 (79)
Diarrhea (Gastrointestinal disorders) | 39 (67)
Fatigue (General disorders) | 51 (111)
Infection (Infections and infestations) | 56 (136)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-10-05): https://cdn.clinicaltrials.gov/large-docs/71/NCT01816971/Prot_SAP_000.pdf
  • Informed Consent Form (2018-05-04): https://cdn.clinicaltrials.gov/large-docs/71/NCT01816971/ICF_001.pdf